CLINICAL TRIAL: NCT01451489
Title: A Randomized,Multicentre,Prospective Study on the Tacrolimus(FK506)for Focal Segmental Glomerulosclerosis
Brief Title: The Efficacy and Safety of Tacrolimus in Treated Refractory Focal Segmental Glomerulosclerosis
Acronym: FSGS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment of subject is very difficult
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhi-Hong Liu, M.D., Professor, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-1101
Record Dates: First submitted 2011-08-05; First posted 2011-10-13 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: FSGS
Keywords: FSGS; FK506; CTX
MeSH Terms: interventions — Tacrolimus; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclophosphamide (Active Comparator): CTX
  Interventions: Drug: Cyclophosphamide
- FK506 (Experimental): 0.05-0.1mg/kg/d;adjust the dose according the serum concentration(aim 5-10ng/ml),maximum dose 6mg/day;divided in twice, interval 12 hours.
  Interventions: Drug: FK506

INTERVENTIONS:
Drug: FK506 — FK506:0.05-0.1mg/kg/d
  Other Names: Tacrolimus,Prograf
  Arms: FK506
Drug: Cyclophosphamide — CTX 750mg/m2 per month in the induction phase,then 750mg/m2 every 2 month for 3 times,then 750mg/m2 every 3 months.
  Other Names: CTX
  Arms: Cyclophosphamide

SUMMARY:
This is a prospective,multicentre study to compare the efficacy, safety, tolerability and relapse of FK506 versus CTX in the treatment of severe Focal Segmental Glomerulosclerosis (FSGS).

DETAILED DESCRIPTION:
1. Using the response rate and completely response time to compare the efficacy of FK506 versus CTX therapy for the severe FSGS patients.
2. To compare the safety and tolerability of FK506 versus CTX for the severe FSGS patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of FSGS.
* Patients with a proteinuria ≥ 3.5g/24h,and blood albumin <30g/L,and Scr< 2.3 mg/dl and eGFR>30ml/min per 1.73m2.
* Patients who signed written informed consent form (patients less than 18 years old with their parents/legal representative's signatures), and have given their consent to follow all study procedures and follow-up.

Exclusion Criteria:

* Patients who have received treatment of FK506 in latest 2 month or the cumulative dose CTX≥6 g.
* Patients who are known to be allergic to a macrolide.
* Patients who have active hepatitis.
* Patients who have impaired liver function, with ALT/GPT or AST/GOT twice more than the normal upper limit .
* Patients with blood leukocyte < 3000/ul.
* Patients with kidney disease family history
* Patients with 2 type diabetes.
* Patients with obesity whose BMI>28kg/m2.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-10-13 (Actual); Primary Completion 2016-03-23 (Actual); Study Completion 2016-10-29 (Actual)

PRIMARY OUTCOMES:
the rates of the complete remission during the induction phase | 6 months

SECONDARY OUTCOMES:
the total remission rates | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, MD, Study Director — Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine
Locations (1):
- Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Hodson EM, Sinha A, Cooper TE. Interventions for focal segmental glomerulosclerosis in adults. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD003233. doi: 10.1002/14651858.CD003233.pub3. PMID 35224732